CLINICAL TRIAL: NCT00702845
Title: A Phase III, Randomized, Double-blind, Active-controlled, Equivalence Clinical Trial to Investigate the Efficacy and Safety of a Single Injection of 100 µg Org 36286 (Corifollitropin Alfa) to Induce Multifollicular Development for Controlled Ovarian Stimulation (COS) Using Daily Recombinant FSH (recFSH) as a Reference
Brief Title: To Investigate Efficacy and Safety of a Single Injection of Org 36286 for Ovarian Stimulation Using Daily Recombinant FSH as Reference (Ensure)(P05690/MK-8962-001)
Acronym: Ensure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P05690; 2006-003811-36 (EudraCT Number); 107012 (Other: Organon Study Number)
Record Dates: First submitted 2008-06-18; First posted 2008-06-20 (Estimated); Results first posted 2015-04-27 (Estimated); Last update posted 2024-06-18 (Actual); Status verified 2022-02

CONDITIONS: Infertility
Keywords: In vitro fertilization; Pharmacological effects of drugs; Hormones; Hormone Substitutes and Hormone Antagonists; Pharmacological Actions; Randomized; Multi-center; Multi-national; Double-blind; Active-controlled; Equivalence
MeSH Terms: conditions — Infertility | interventions — follicle stimulating hormone, human, with HCG C-terminal peptide; follitropin beta; Glycoprotein Hormones, alpha Subunit; Gonadotropin-Releasing Hormone; ganirelix; Progesterone; follitropin alfa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- corifollitropin alfa 100 µg (Experimental): Participants received a single subcutaneous (SC) injection of corifollitropin alfa 100 μg (Org 36286) on Day 2 or 3 of the menstrual cycle and daily placebo-recombinant Follicle Stimulating Hormone (recFSH) injections (7 total) from Stimulation Day 1 up to and including Stimulation Day 7. Participants also received open-label recFSH (up to 200 IU/day) from Stimulation Day 8 onwards, up to and including Day of Human Chorion Gonadotropin (hCG) administration. Participants also received Gonadotropin Releasing Hormone (GnRH) antagonist ganirelix (0.25 mg) once daily SC starting on Stimulation Day 5 up to and including the Day of hCG (10,000 or 5,000 IU/USP). Participants also received progesterone (at least 600 mg/day vaginally or 50 mg/day by intramuscular [IM] injection), starting on day of oocyte pick-up (OPU) and continuing for at least 6 weeks or up to menses.
  Interventions: Drug: corifollitropin alfa (Org 36286); Drug: gonadatropin releasing hormone (GnRH) antagonist (ganirelix); Drug: human chorion gonadatropin (hCG); Biological: progesterone; Drug: placebo-recFSH (follitropin alfa); Biological: open-label recFSH
- recFSH 150 IU (Active Comparator): Participants in the reference group received a single SC injection of placebo-corifollitropin alfa administered on Day 2 or 3 of the menstrual cycle and daily SC recFSH 150 IU injections (7 total) from Stimulation Day 1 up to and including Stimulation Day 7. Participants also received open-label recFSH (up to 200 IU/day) from Stimulation Day 8 onwards, up to and including the day of hCG (10,000 or 5,000 IU/USP) administration. Participants also received the GnRH antagonist ganirelix (0.25 mg) once daily SC starting on Stimulation Day 5 up to and including the Day of hCG. Participants also received progesterone (at least 600 mg/day vaginally or 50 mg/day IM), starting on the day of OPU and continuing for at least 6 weeks or up to menses.
  Interventions: Drug: recFSH (follitropin beta); Drug: gonadatropin releasing hormone (GnRH) antagonist (ganirelix); Drug: human chorion gonadatropin (hCG); Biological: progesterone; Drug: placebo-corifollitropin alfa; Biological: open-label recFSH

INTERVENTIONS:
Drug: corifollitropin alfa (Org 36286) — 100 µg corifollitropin alfa subcutaneous (SC) injection
  Other Names: Org 36286
  Arms: corifollitropin alfa 100 µg
Drug: recFSH (follitropin beta) — 150 IU recFSH SC injection
  Other Names: recFSH (Puregon/Follistim AQ Cartridge)
  Arms: recFSH 150 IU
Drug: gonadatropin releasing hormone (GnRH) antagonist (ganirelix) — GnRH antagonist (ganirelix) administered SC at a dose of 0.25 mg/day
Drug: human chorion gonadatropin (hCG) — hCG 5,000 IU or 10,000 IU administered SC
Biological: progesterone — Progesterone was started on the day of oocyte pick-up (OPU) and continued for at least 6 weeks or up to menses. Participants received at least 600 mg/day vaginally or 50 mg/day IM.
Drug: placebo-recFSH (follitropin alfa) — Placebo-recFSH administered at the equivalent volume of 150 IU/day.
  Arms: corifollitropin alfa 100 µg
Drug: placebo-corifollitropin alfa — Single SC injection of placebo-corifollitropin alfa administered on Day 2 or 3 of the menstrual cycle.
  Arms: recFSH 150 IU
Biological: open-label recFSH — Open-label recFSH administered up to a maximum dose of 200 IU/day.

SUMMARY:
Clinical trial objectives are to investigate the efficacy and safety of a single injection of 100 μg Org 36286 in women weighing 60 kg or less to induce multifollicular development for controlled ovarian stimulation (COS), using daily recFSH as a reference.

DETAILED DESCRIPTION:
This is a randomized, double-blind, active-controlled, equivalence clinical trial investigating the efficacy and safety of a new treatment regimen with Org 36286, a recombinant gonadotropin applied to initiate and sustain follicular stimulation in COS for Assisted Reproductive Technology (ART). For this regimen, patients receive a single injection of Org 36286 and one week later, treatment is continued with daily recFSH up to the day of triggering final oocyte maturation. In the reference group patients receive daily injections of recFSH up to the day of triggering final oocyte maturation. Equivalence between the two treatment groups in the number of oocytes retrieved is the primary objective of this trial.

ELIGIBILITY:
Inclusion Criteria:

* Females of couples with an indication for COS and IVF or ICSI;
* >=18 and <= 36 years of age at the time of signing informed consent;
* Body weight <= 60 kg and BMI >= 18 and <= 32 kg/m^2;
* Normal menstrual cycle length: 24-35 days;
* Availability of ejaculatory sperm (use of donated and/or cryopreserved sperm is allowed);
* Willing and able to sign informed consent.

Exclusion Criteria:

* History of/or any current (treated) endocrine abnormality;
* History of ovarian hyper-response or ovarian hyperstimulation syndrome

(OHSS);

* History of/or current polycystic ovary syndrome (PCOS);
* More than 20 basal antral follicles <11 mm (both ovaries combined) as measured on USS in the early follicular phase (menstrual cycle day 2-5);
* Less than 2 ovaries or any other ovarian abnormality (including endometrioma > 10 mm; visible on USS);
* Presence of unilateral or bilateral hydrosalphinx (visible on USS);
* Presence of any clinically relevant pathology affecting the uterine cavity or fibroids >= 5 cm;
* More than three unsuccessful IVF cycles since the last established ongoing

pregnancy (if applicable);

* History of non- or low ovarian response to FSH/hMG treatment;
* History of recurrent miscarriage (3 or more, even when unexplained);
* FSH > 12 IU/L or LH > 12 IU/L as measured by the local laboratory (sample taken during the early follicular phase: menstrual cycle day 2-5);
* Any clinically relevant abnormal laboratory value based on a sample taken during the screening phase;
* Contraindications for the use of gonadotropins (e.g. tumors, pregnancy/lactation, undiagnosed vaginal bleeding, hypersensitivity, ovarian cysts);
* Recent history of/or current epilepsy, HIV infection, diabetes, cardiovascular,

gastro-intestinal, hepatic, renal or pulmonary disease;

* Abnormal karyotyping of the patient or her partner (if karyotyping is performed);
* Smoking more than 5 cigarettes per day;
* History or presence of alcohol or drug abuse within 12 months prior to signing informed consent;
* Previous use of Org 36286;
* Use of hormonal preparations within 1 month prior to randomization;
* Hypersensitivity to any of the concomitant medication prescribed as part of the treatment regimen in this protocol;
* Administration of investigational drugs within three months prior to signing informed consent.

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 397 (Actual)
Dates: Start 2006-12-28 (Actual); Primary Completion 2007-07-07 (Actual); Study Completion 2007-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Corifollitropin alfa Ensure Study Group. Corifollitropin alfa for ovarian stimulation in IVF: a randomized trial in lower-body-weight women. Reprod Biomed Online. 2010 Jul;21(1):66-76. doi: 10.1016/j.rbmo.2010.03.019. Epub 2010 Mar 28. PMID 20483664
- [Derived] Zandvliet AS, Prohn M, de Greef R, van Aarle F, McCrary Sisk C, Stegmann BJ. Impact of patient characteristics on the pharmacokinetics of corifollitropin alfa during controlled ovarian stimulation. Br J Clin Pharmacol. 2016 Jul;82(1):74-82. doi: 10.1111/bcp.12939. Epub 2016 May 31. PMID 26991902
- [Derived] Griesinger G, Verweij PJ, Gates D, Devroey P, Gordon K, Stegmann BJ, Tarlatzis BC. Prediction of Ovarian Hyperstimulation Syndrome in Patients Treated with Corifollitropin alfa or rFSH in a GnRH Antagonist Protocol. PLoS One. 2016 Mar 7;11(3):e0149615. doi: 10.1371/journal.pone.0149615. eCollection 2016. PMID 26950065

RESULTS

PARTICIPANT FLOW:
Groups:
- 100 μg Corifollitropin Alfa: Participants received a single subcutaneous (SC) injection of corifollitropin alfa 100 μg (Org 36286) on Day 2 or 3 of the menstrual cycle and daily placebo-recombinant Follicle Stimulating Hormone (recFSH) injections (7 total) from Stimulation Day 1 up to and including Stimulation Day 7. Participants also received open-label recFSH (up to 200 IU/day) from Stimulation Day 8 onwards, up to and including Day of Human Chorion Gonadotropin (hCG) administration. Participants also received Gonadotropin Releasing Hormone (GnRH) antagonist ganirelix (0.25 mg) once daily SC starting on Stimulation Day 5 up to and including the Day of hCG (10,000 or 5,000 IU/USP). Participants also received progesterone (at least 600 mg/day vaginally or 50 mg/day by intramuscular [IM] injection), starting on day of oocyte pick-up (OPU) and continuing for at least 6 weeks or up to menses.
- 150 IU recFSH: Participants received a single SC injection of placebo-corifollitropin alfa administered on Day 2 or 3 of the menstrual cycle and daily SC recFSH 150 IU injections (7 total) from Stimulation Day 1 up to and including Stimulation Day 7. Participants also received open-label recFSH (up to 200 IU/day) from Stimulation Day 8 onwards, up to and including the day of hCG (10,000 or 5,000 IU/USP) administration. Participants also received the GnRH antagonist ganirelix (0.25 mg) once daily SC starting on Stimulation Day 5 up to and including the Day of hCG. Participants also received progesterone (at least 600 mg/day vaginally or 50 mg/day IM), starting on the day of OPU and continuing for at least 6 weeks or up to menses.
Period: Overall Study
Arm/Group | 100 μg Corifollitropin Alfa | 150 IU recFSH
Started | 268 | 129 (Includes one treated participant who was not randomized)
Randomized | 268 | 128
Completed | 246 | 121
Not Completed | 22 | 8
Not completed — No/too few/bad quality oocytes retrieved | 2 | 2
Not completed — Too high ovarian response | 5 | 1
Not completed — Risk of ovarian hyperstimulation synd. | 1 | 0
Not completed — Insufficient ovarian response | 1 | 0
Not completed — No/too few/bad quality embryos retrieved | 7 | 1
Not completed — No or abnormal fertilization | 4 | 2
Not completed — Patient's decision | 2 | 1
Not completed — Not randomized | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat group, which consisted of all randomized participants who received corifollitropin alfa or recFSH.
Groups:
- 100 μg Corifollitropin Alfa: Participants received a single SC injection of corifollitropin alfa 100 μg (Org 36286) on Day 2 or 3 of the menstrual cycle and daily placebo-recFSH injections (7 total) from Stimulation Day 1 up to and including Stimulation Day 7. Participants also received open-label recFSH (up to 200 IU/day) from Stimulation Day 8 onwards, up to and including Day of hCG administration. Participants also received GnRH antagonist ganirelix (0.25 mg) once daily SC starting on Stimulation Day 5 up to and including the Day of hCG (10,000 or 5,000 IU/USP). Participants also received progesterone (at least 600 mg/day vaginally or 50 mg/day IM), starting on day of OPU and continuing for at least 6 weeks or up to menses.
- Total: Total of all reporting groups
Arm/Group | 100 μg Corifollitropin Alfa | 150 IU recFSH | Total
Number analyzed (Participants) | 268 | 128 | 396
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.9 (3.2) | 31.1 (3.0) | 31.0 (3.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 268 | 128 | 396
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Cumulus-oocyte-complexes Retrieved, Per Attempt
Description: The primary efficacy parameter was defined as the number of cumulus-oocyte-complexes retrieved from participants in a controlled ovarian stimulation (COS) cycle for in vitro fertilization (IVF) and/or intracytoplasmic sperm injection (ICSI). For participants who did not have cumulus-oocyte-complex retrieval, the number retrieved was set to zero.
Time Frame: One COS cycle with cumulus-oocyte-complex retrieval (up to a maximum total duration of 21 days)
Population: Intent-to-Treat (ITT) Group, which consisted of all randomized participants who received corifollitropin alfa or recFSH.
Measure: Mean (Standard Deviation); unit: Number of cumulus-oocyte-complexes
Arm/Group | 100 μg Corifollitropin Alfa | 150 IU recFSH
Number analyzed (Participants) | 268 | 128
Number of cumulus-oocyte-complexes | 13.3 (7.3) | 10.6 (5.9)
Statistical Analysis 1: Comparison: 100 μg Corifollitropin Alfa vs 150 IU recFSH; Test type: Non-Inferiority or Equivalence — Equivalence margins of -3 and +5 were applied for the difference in the mean number of oocytes between the treatment groups. Org 36286 treatment was considered equivalent to the reference treatment (recFSH) if the two-sided 95% confidence interval of the difference was between -3 and +5 oocytes; p < 0.001, ANOVA; Mean Difference (Final Values) = 2.5, 95% CI 2-sided [1.2 to 3.9]

2. Secondary Outcome: Total Dose of recFSH Administered
Description: Total dose of recFSH (IU) administered was defined as the total amount of recFSH needed by participants to reach the criterion for administration of hCG (at least 3 follicles >=17mm).
Time Frame: One COS cycle (up to a maximum total duration of 19 stimulation days)
Population: Participants from the ITT Group (consisting of all randomized participants who received corifollitropin alfa or recFSH) who received hCG.
Measure: Median (Full Range); unit: International Unit (IU)
Arm/Group | 100 μg Corifollitropin Alfa | 150 IU recFSH
Number analyzed (Participants) | 266 | 127
International Unit (IU) | 300.0 [0 to 1550] | 1350.0 [825 to 2650]

3. Secondary Outcome: Total Dose of recFSH Administered From Day 8 Onwards
Description: Total dose of recFSH (IU) needed from Stimulation Day 8 onwards to reach the criterion for administration of hCG (at least 3 follicles >=17mm).
Time Frame: Stimulation Day 8 of COS cycle up to day of hCG administration (up to a maximum total duration of 19 stimulation days)
Population: as for outcome 2
Measure: Median (Full Range); unit: International Unit (IU)
Arm/Group | 100 μg Corifollitropin Alfa | 150 IU recFSH
Number analyzed (Participants) | 266 | 127
International Unit (IU) | 300.0 [0 to 1550] | 275.0 [0 to 1600]

4. Secondary Outcome: Number of Days Treated With recFSH
Description: Numbers of days treated with recFSH was defined as the total number of days participants received recFSH (excluding coasting days) until they reached the criterion for administration of hCG (at least 3 follicles >=17mm).
Time Frame: One COS cycle (up to a maximum total duration of 19 stimulation days)
Population: as for outcome 2
Measure: Median (Full Range); unit: Days
Arm/Group | 100 μg Corifollitropin Alfa | 150 IU recFSH
Number analyzed (Participants) | 266 | 127
Days | 2.0 [0 to 7] | 9.0 [6 to 15]

5. Secondary Outcome: Total Duration of Stimulation (Days)
Description: Total duration of stimulation was defined as the number of days from first drug administration up to and including the Day of hCG administration.
Time Frame: One COS cycle (up to a maximum total duration of 19 stimulation days)
Population: as for outcome 2
Measure: Median (Full Range); unit: Days
Arm/Group | 100 μg Corifollitropin Alfa | 150 IU recFSH
Number analyzed (Participants) | 266 | 127
Days | 9.0 [6 to 15] | 9.0 [6 to 15]

6. Secondary Outcome: Serum Follicle Stimulating Hormone (FSH) Levels (Restricted to Participants With hCG Injection)
Description: Blood samples for assessment of serum FSH were taken prior to injection on Stimulation Day 1, Day 3, Day 5, Day 8, Day of hCG, Day of ET, at the visit two weeks after ET.
Time Frame: Predose up to 2 weeks after ET (up to maximum of 6 weeks)
Population: as for outcome 2
Measure: Median (Full Range); unit: IU/L
Arm/Group | 100 μg Corifollitropin Alfa | 150 IU recFSH
Number analyzed (Participants) | 268 | 127
IU/L
  Stimulation Day 1 (pre-dose) (n=265,122) | 6.46 (1.84) [1.2 to 14.0] | 6.51 (1.89) [1.9 to 15.4]
  Stimulation Day 3 (n=265,127) | 26.30 (7.14) [15.2 to 51.1] | 9.18 (2.48) [4.7 to 22.3]
  Stimulation Day 5 (n=265,127) | 19.50 (4.52) [0.8 to 34.7] | 10.20 (2.98) [1.0 to 28.0]
  Stimulation Day 8 (n=255,121) | 10.10 (2.12) [5.0 to 18.1] | 10.30 (2.26) [4.5 to 23.6]
  Day of hCG injection (n=262,126) | 11.50 (2.65) [5.0 to 19.9] | 10.65 (3.57) [5.9 to 41.8]
  Day of ET (n=242,121) | 2.52 (1.05) [0.4 to 5.8] | 1.32 (1.02) [0.4 to 8.4]
  2 weeks after ET (n=245,121) | 4.46 (3.53) [0.1 to 16.6] | 1.90 (NA) [0.1 to 11.5]

7. Secondary Outcome: Serum Lutenizing Hormone (LH) Levels (Restricted to Participants With hCG Injection)
Description: Blood samples for assessment of serum LH were taken prior to injection on Stimulation Day 1, Day 3, Day 5, Day 8, Day of hCG, Day of ET, at the visit two weeks after ET.
Time Frame: Predose up to 2 weeks after ET (up to maximum of 6 weeks)
Population: as for outcome 2
Measure: Median (Full Range); unit: IU/L
Arm/Group | 100 μg Corifollitropin Alfa | 150 IU recFSH
Number analyzed (Participants) | 266 | 127
IU/L
  Stimulation Day 1 (pre-dose) (n=265,122) | 4.46 (1.81) [0.3 to 13.3] | 4.12 (1.94) [0.3 to 14.7]
  Stimulation Day 3 (n=265,127) | 1.18 (0.80) [0.3 to 6.3] | 1.46 (1.00) [0.3 to 6.8]
  Stimulation Day 5 (n=264,127) | 1.91 (3.70) [0.3 to 33.3] | 1.49 (7.26) [0.3 to 76.7]
  Stimulation Day 8 (n=255,121) | 0.82 (NA) [0.3 to 9.9] | 1.60 (2.35) [0.3 to 17.8]
  Day of hCG injection (n=262,126) | 0.88 (NA) [0.3 to 9.9] | 1.30 (2.06) [0.3 to 12.5]
  Day of ET (n=242,121) | NA (NA) [0.3 to 4.1] — If more than 1/2 of the values per assessment day were smaller than the lower limit of quantification (LLOQ) (0.6 IU/L), the median was reported as missing. | NA (NA) [0.3 to 5.6] — If more than 1/2 of the values per assessment day were smaller than LLOQ (0.6 IU/L), the median was reported as missing.
  2 weeks after ET (n=245,121) | 2.38 (NA) [0.3 to 16.2] | 1.02 (NA) [0.3 to 24.4]

8. Secondary Outcome: Serum Estradiol (E2) Levels (Restricted to Participants With hCG Injection)
Description: Blood samples for assessment of serum E2 were taken prior to injection on Stimulation Day 1, Day 3, Day 5, Day 8, Day of hCG, Day of ET, at the visit two weeks after ET.
Time Frame: Predose up to 2 weeks after ET (up to maximum of 6 weeks)
Population: as for outcome 2
Measure: Median (Full Range); unit: pmol/L
Arm/Group | 100 μg Corifollitropin Alfa | 150 IU recFSH
Number analyzed (Participants) | 266 | 127
pmol/L
  Stimulation Day 1 (pre-dose) (n=265,122) | 118.17 (53.18) [25.0 to 466.1] | 120.38 (71.07) [25.0 to 748.7]
  Stimulation Day 3 (n=265,127) | 803.73 (553.18) [76.7 to 4917.8] | 506.46 (369.66) [25.0 to 2719.5]
  Stimulation Day 5 (n=265,127) | 1901.06 (1490.48) [165.9 to 9578.7] | 1295.51 (1015.75) [25.0 to 6128.9]
  Stimulation Day 8 (n=255,121) | 2899.30 (2632.83) [282.2 to 20441.9] | 3167.21 (2710.16) [111.2 to 14606.6]
  Day of hCG injection (n=262,126) | 4440.70 (3355.95) [690.0 to 20441.9] | 4440.70 (3114.93) [987.2 to 16111.3]
  Day of ET (n=242,121) | 3475.49 (2640.49) [433.1 to 16258.1] | 3670.00 (2946.26) [612.9 to 18460.1]
  2 weeks after ET (n=245,121) | 168.45 (3002.09) [25.0 to 17579.3] | 392.69 (2889.61) [25.0 to 18313.3]

9. Secondary Outcome: Serum Progesterone (P) Levels (Restricted to Participants With hCG Injection)
Description: Blood samples for assessment of serum P were taken prior to injection on Stimulation Day 1, Day 3, Day 5, Day 8, Day of hCG, Day of ET, at the visit two weeks after ET.
Time Frame: Predose up to 2 weeks after ET (up to maximum of 6 weeks)
Population: as for outcome 2
Measure: Median (Full Range); unit: nmol/L
Arm/Group | 100 μg Corifollitropin Alfa | 150 IU recFSH
Number analyzed (Participants) | 266 | 127
nmol/L
  Stimulation Day 1 (pre-dose) (n=264,120) | 1.36 (2.90) [0.6 to 33.4] | 1.40 (0.97) [0.6 to 9.3]
  Stimulation Day 3 (n=263,126) | 1.23 (NA) [0.6 to 11.7] | NA (NA) [0.6 to 3.3] — If more than 1/2 of the values per assessment day were smaller than LLOQ (1.2 nmol/L), the median was reported as missing.
  Stimulation Day 5 (n=265,127) | 1.65 (3.27) [0.6 to 53.7] | 1.28 (NA) [0.6 to 93.8]
  Stimulation Day 8 (n=255,121) | 1.39 (0.64) [0.6 to 3.3] | 2.03 (1.11) [0.6 to 6.2]
  Day of hCG injection (n=262,126) | 2.10 (1.34) [0.6 to 8.4] | 2.39 (1.78) [0.6 to 15.6]
  Day of ET (n=242,121) | 421.35 (223.93) [82.7 to 960.4] | 333.90 (157.38) [45.2 to 852.2]
  2 weeks after ET (n=244,120) | 38.64 (263.88) [0.6 to 960.4] | 51.99 (236.91) [0.6 to 960.4]

10. Secondary Outcome: Serum Inhibin-B Levels (Restricted to Participants With hCG Injection)
Description: Blood samples for assessment of serum inhibin-B were taken prior to injection on Stimulation Day 1, Day 3, Day 5, Day 8, Day of hCG, Day of ET, at the visit two weeks after ET.
Time Frame: Predose up to 2 weeks after ET (up to maximum of 6 weeks)
Population: as for outcome 2
Measure: Median (Full Range); unit: pg/mL
Arm/Group | 100 μg Corifollitropin Alfa | 150 IU recFSH
Number analyzed (Participants) | 266 | 127
pg/mL
  Stimulation Day 1 (pre-dose) (n=265,123) | 54.20 (26.40) [5.0 to 178.0] | 57.80 (168.69) [5.0 to 1910.0]
  Stimulation Day 3 (n=265,127) | 351.00 (216.79) [5.0 to 1590.0] | 259.00 (143.21) [5.0 to 747.0]
  Stimulation Day 5 (n=264,127) | 598.00 (527.96) [17.3 to 3080.0] | 489.00 (348.64) [5.0 to 2470.0]
  Stimulation Day 8 (n=255,121) | 619.00 (643.76) [56.0 to 4000.0] | 650.00 (536.39) [20.1 to 2670.0]
  Day of hCG injection (n=262,126) | 729.50 (721.20) [56.0 to 4000.0] | 615.50 (571.49) [5.0 to 2870.0]
  Day of ET (n=242,121) | 18.20 (25.49) [5.0 to 173.0] | 17.00 (29.36) [5.0 to 167.0]
  2 weeks after ET (n=245,121) | 17.50 (NA) [5.0 to 613.0] | NA (NA) [5.0 to 163.0] — If more than 1/2 of the values per assessment day were smaller than LLOQ (10 pg/mL), the median was reported as missing

11. Secondary Outcome: Number and Size Distribution of Follicles During Stimulation and on the Day of hCG Administration
Description: For each participant, the number of follicles ≥11 mm, ≥15 mm, and ≥17 mm, documented by ultrasonography on defined days during the treatment cycle, was calculated.
Time Frame: Predose up to day of hCG administration (up to a maximum total duration of 19 stimulation days, including day of hCG administration)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Follicles
Arm/Group | 100 μg Corifollitropin Alfa | 150 IU recFSH
Number analyzed (Participants) | 268 | 128
Follicles
  Stimulation Day 1, >=11mm (n=266,124) | 0.0 (0.1) | 0.0 (0.2)
  Stimulation Day 1, >=15mm (n=266,124) | 0.0 (0.1) | 0.0 (0.0)
  Stimulation Day 1, >=17mm (n=266,124) | 0.0 (0.1) | 0.0 (0.0)
  Stimulation Day 3, >=11mm (n=268,128) | 0.6 (1.7) | 0.5 (0.9)
  Stimulation Day 3, >=15mm (n=268,128) | 0.0 (0.1) | 0.0 (0.0)
  Stimulation Day 3, >=17mm (n=268,128) | 0.0 (0.0) | 0.0 (0.0)
  Stimulation Day 5, >=11mm (n=267,128) | 4.7 (3.6) | 4.1 (3.2)
  Stimulation Day 5, >=15mm (n=267,128) | 0.3 (0.7) | 0.3 (0.9)
  Stimulation Day 5, >=17mm (n=267,128) | 0.0 (0.2) | 0.0 (0.1)
  Stimulation Day 6, >=11mm (n=9,5) | 7.6 (5.2) | 8.6 (6.3)
  Stimulation Day 6, >=15mm (n=9,5) | 1.8 (3.0) | 4.0 (3.8)
  Stimulation Day 6, >=17mm (n=9,5) | 0.7 (1.3) | 1.8 (2.0)
  Stimulation Day 7, >=11mm (n=30,12) | 11.9 (6.8) | 9.2 (4.4)
  Stimulation Day 7, >=15mm (n=30,12) | 4.5 (4.7) | 3.3 (2.8)
  Stimulation Day 7, >=17mm (n=30,12) | 1.8 (2.8) | 1.1 (1.3)
  Stimulation Day 8, >=11mm (n=259,121) | 11.8 (6.1) | 10.6 (5.3)
  Stimulation Day 8, >=15mm (n=259,121) | 5.0 (4.6) | 5.1 (4.5)
  Stimulation Day 8, >=17mm (n=259,121) | 2.0 (3.0) | 2.4 (3.1)
  Stimulation Day 9, >=11mm (n=185,76) | 13.4 (6.5) | 11.1 (5.0)
  Stimulation Day 9, >=15mm (n=185,76) | 6.9 (4.7) | 6.0 (4.5)
  Stimulation Day 9, >=17mm (n=185,76) | 2.6 (2.5) | 2.6 (2.5)
  Stimulation Day 10, >=11mm (n=101,40) | 13.9 (6.7) | 13.0 (6.4)
  Stimulation Day 10, >=15mm (n=101,40) | 7.4 (4.9) | 7.5 (5.3)
  Stimulation Day 10, >=17mm (n=101,40) | 3.6 (3.5) | 4.0 (4.0)
  Stimulation Day 11, >=11mm (n=38,14) | 13.9 (6.7) | 11.6 (7.1)
  Stimulation Day 11, >=15mm (n=38,14) | 7.7 (5.7) | 7.1 (4.6)
  Stimulation Day 11, >=17mm (n=38,14) | 3.9 (3.8) | 3.8 (3.5)
  Stimulation Day 12, >=11mm (n=17,6) | 12.7 (5.4) | 9.3 (4.0)
  Stimulation Day 12, >=15mm (n=17,6) | 6.8 (3.5) | 5.2 (2.9)
  Stimulation Day 12, >=17mm (n=17,6) | 3.5 (2.8) | 2.7 (2.1)
  Stimulation Day 13, >=11mm (n=5,4) | 17.0 (9.5) | 10.3 (5.4)
  Stimulation Day 13, >=15mm (n=5,4) | 10.6 (8.6) | 6.3 (4.5)
  Stimulation Day 13, >=17mm (n=5,4) | 4.4 (6.2) | 4.0 (3.4)
  Stimulation Day 14, >=11mm (n=2,1) | 13.5 (12.0) | 3.0 (0.0)
  Stimulation Day 14, >=15mm (n=2,1) | 10.5 (12.0) | 0.0 (0.0)
  Stimulation Day 14, >=17mm (n=2,1) | 6.0 (5.7) | 0.0 (0.0)
  Stimulation Day 15, >=11mm (n=1,1) | 7.0 (0.0) | 4.0 (0.0)
  Stimulation Day 15, >=15mm (n=1,1) | 4.0 (0.0) | 4.0 (0.0)
  Stimulation Day 15, >=17mm (n=1,1) | 2.0 (0.0) | 3.0 (0.0)
  Day of hCG administration, >=11mm (n=266,127) | 14.9 (6.6) | 12.9 (5.8)
  Day of hCG administration, >=15mm (n=266,127) | 9.4 (4.9) | 8.5 (4.4)
  Day of hCG administration, >=17mm (n=266,127) | 5.3 (3.0) | 5.1 (3.0)

12. Secondary Outcome: Number and Quality of Oocytes Assessed Prior to ICSI (Restricted to Participants With ICSI Only)
Description: The number of oocytes used for ICSI was assessed and categorized based on their quality (i.e., metaphase I oocytes, metaphase II oocytes, and germinal vesicles stage oocytes).
Time Frame: Up to 36 hours after administration of hCG
Population: Participants from the ITT Group (consisting of all randomized participants who received corifollitropin alfa or recFSH) who underwent ICSI.
Measure: Mean (Standard Deviation); unit: Number of oocytes
Arm/Group | 100 μg Corifollitropin Alfa | 150 IU recFSH
Number analyzed (Participants) | 137 | 72
Number of oocytes
  Oocytes assessed prior to ICSI | 12.7 (6.8) | 9.9 (5.4)
  Metaphase I oocytes | 0.8 (1.2) | 0.7 (1.2)
  Metaphase II oocytes | 10.7 (6.4) | 7.8 (4.8)
  Germinal vesicles stage oocytes | 1.1 (1.6) | 1.3 (2.1)

13. Secondary Outcome: Fertilization Rate
Description: Fertilization rate, defined as 100 times the ratio of the number of fertilized 2 pronuclei (PN) oocytes obtained and the number of oocytes incubated, was tabulated for each treatment group.
Time Frame: Up to 10 weeks after ET
Population: Participants from the ITT Group (consisting of all randomized participants who received corifollitropin alfa or recFSH) who received fertilized oocytes.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | 100 μg Corifollitropin Alfa | 150 IU recFSH
Number analyzed (Participants) | 264 | 124
Percentage | 67.6 (22.5) | 67.7 (25.4)

14. Secondary Outcome: Number and Quality of Embryos Obtained at Day 3 (Restricted to Participants With IVF and/or ICSI)
Description: Embryo quality was rated Grade 1, 2, 3, or other. Grade 1 represented excellent quality; Grade 2 good quality; Grade 3 fair quality. "Other" grade embryos were those that did not qualify as Grade 1, 2, or 3.
Time Frame: Post fertilization Day 3 (up to a maximum of 2 days after hCG administration)
Population: Participants from the ITT Group (consisting of all randomized participants who received corifollitropin alfa or recFSH) who underwent IVF and/or ICSI.
Measure: Mean (Standard Deviation); unit: Number of embryos
Arm/Group | 100 μg Corifollitropin Alfa | 150 IU recFSH
Number analyzed (Participants) | 264 | 124
Number of embryos
  Total (n=259,123) | 7.2 (4.1) | 6.2 (4.0)
  Good quality | 3.4 (3.0) | 3.0 (3.0)
  Grade 1 | 1.7 (2.3) | 1.4 (2.1)
  Grade 2 | 1.8 (1.9) | 1.6 (1.9)
  Grade 3 | 2.8 (2.8) | 2.4 (2.4)
  Other | 1.0 (1.6) | 0.7 (1.7)

15. Secondary Outcome: Implantation Rate for Participants With ET
Description: The implantation rate was defined as 100 times the maximum number of gestational sacs as assessed by any ultrasound scan (USS) after ET divided by the number of embryos transferred (per participant), maximized to 100%.
Time Frame: Up to 6 weeks after ET within a treatment cycle (up to a maximum 10 weeks)
Population: Participants from the ITT Group (consisting of all randomized participants who received corifollitropin alfa or recFSH) who underwent ET.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | 100 μg Corifollitropin Alfa | 150 IU recFSH
Number analyzed (Participants) | 246 | 121
Percentage | 23.6 (37.4) | 28.5 (38.6)

16. Secondary Outcome: Number of Participants With Miscarriages
Description: A miscarriage, also known as a "spontaneous abortion," was defined as the loss of a fetus without induction or instrumentation.
Time Frame: Up to 10 weeks after ET (up to a maximum of 14 weeks)
Population: Participants from the ITT Group (consisting of all randomized participants who received corifollitropin alfa or recFSH) who had a biological pregnancy.
Measure: Number; unit: Participants
Arm/Group | 100 μg Corifollitropin Alfa | 150 IU recFSH
Number analyzed (Participants) | 268 | 128
Participants
  Per clinical pregnancy (n=78,48) | 10 (12.8) | 4 (8.3)
  Per vital pregnancy (n=69,45) | 1 | 1

17. Secondary Outcome: Number of Participants With Pregnancies
Description: A Biochemical Pregnancy was defined as a pregnancy proven by a biochemical pregnancy test. (Participants not having a positive biochemical pregnancy test result, but with an ultrasound showing at least one gestational sac were counted as having a biochemical pregnancy.) A Clinical Pregnancy was defined as the presence of at least one gestational sac as assessed by an USS scan. A Vital Pregnancy was considered the presence of at least one fetus with heart activity as assessed by USS. An Ongoing Pregnancy was defined as the presence of at least one fetus with heart activity at least 10 weeks after ET as assessed by USS or Doppler, or confirmed by live birth.
Time Frame: Up to 10 weeks after ET (up to a maximum of 14 weeks)
Population: ITT Group, which consisted of all randomized participants who received corifollitropin alfa or recFSH.
Measure: Number; unit: Participants
Arm/Group | 100 μg Corifollitropin Alfa | 150 IU recFSH
Number analyzed (Participants) | 268 | 128
Participants
  Biochemical pregnancy, per attempt (n=268,128) | 101 | 58
  Biochemical pregnancy, per ET (n=246,121) | 101 | 58
  Clinical pregnancy, per attempt (n=268,128) | 78 | 48
  Clinical pregnancy, per ET (n=246,121) | 78 | 48
  Vital pregnancy, per attempt (n=268,128) | 69 | 45
  Vital pregnancy, per ET (n=246,121) | 69 | 45
  Ongoing pregnancy, per attempt (n=268,128) | 68 | 44
  Ongoing pregnancy, per ET (n=246,121) | 68 | 44

ADVERSE EVENTS:
Time Frame: Up to 10 weeks after ET (up to a maximum of 14 weeks)
Description: All Participants Treated Group, which included one treated participant who was not randomized.
Arm/Group | 100 μg Corifollitropin Alfa | 150 IU recFSH
Serious Adverse Events (participants affected / at risk) | 20/268 | 9/129
Other Adverse Events (participants affected / at risk) | 107/268 | 55/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 100 μg Corifollitropin Alfa (N=268) | 150 IU recFSH (N=129)
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0)
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Antepartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 8 (8) | 2 (2)
Heterotopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Imminent abortion (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Ruptured ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 7 (7) | 0 (0)
Ovarian torsion (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Abortion induced (Surgical and medical procedures) | 0 (0) | 1 (1)
Selective abortion (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 100 μg Corifollitropin Alfa (N=268) | 150 IU recFSH (N=129)
Nasopharyngitis (Infections and infestations) | 13 (13) | 7 (7)
Headache (Nervous system disorders) | 25 (30) | 12 (17)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 14 (14) | 8 (8)
Antepartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 18 (22) | 17 (17)
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 14 (15) | 6 (7)
Pelvic discomfort (Reproductive system and breast disorders) | 27 (42) | 19 (24)
Pelvic pain (Reproductive system and breast disorders) | 29 (30) | 14 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any scientific paper, presentation, or other communication concerning the clinical trial described in this protocol will first be submitted to the sponsor, at least six weeks ahead of estimated publication or presentation, for written consent, which shall not be withheld unreasonably.